CLINICAL TRIAL: NCT00006419
Title: Diet and Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 935; R01HL063841 (NIH)
Record Dates: First submitted 2000-10-26; First posted 2000-10-27 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-05

CONDITIONS: Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To examine the relationship of specific dietary factors to risk of chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
BACKGROUND:

Although tobacco smoking is the major environmental risk factor for COPD, only a minority of smokers develops this condition, and it appears that genetic and other environmental factors are important in determining risk. There has been growing interest in the hypothesis that dietary factors modify COPD risk, possibly by protecting against oxidant injury. Available data addressing this hypothesis have a variety of methodological limitations that preclude any firm conclusions. The study was the first to address this hypothesis using data from the Nurses' Health Study, a large, prospective cohort study with detailed dietary assessments and a follow-up interval of sufficient duration to examine incident COPD.

DESIGN NARRATIVE:

The study examined the relationship between dietary factors and chronic obstructive pulmonary disease (COPD) among participants in the Nurses' Health Study, an ongoing prospective cohort study of 121,700 women, ages 39-64 in 1985. This cohort had been followed by means of biennial questionnaires which inquired about a variety of topics, including dietary intake (using a validated semi-quantitative food frequency questionnaire) and physician diagnosis of COPD. In 1998, all participants with a history of COPD were sent a supplementary questionnaire regarding specifics of COPD diagnosis and related topics. The study examined the relation of dietary factors to risk of newly-diagnosed COPD during 1985-1998. During this time period, there were approximately 2,100 cases of "confirmed" COPD (i.e., physician diagnosis and pulmonary function tests [PFTs] at time of diagnosis or abnormal FEV-I in past year) and "probable" COPD (i.e., physician diagnosis and recent respiratory symptoms, but PFTs not known). Preliminary data supported the validity of these case definitions, and this was examined further by reviewing 600 medical records. Likewise, potential under-diagnosis was examined in a random sample of past and current smokers who had never reported COPD or asthma. The specific dietary hypotheses were that high intakes of antioxidants (e.g., vitamin C, vitamin E, and carotenoids), magnesium, potassium, and n-3 polyunsaturated fatty acids (e.g., fish oils) decreased risk of COPD, whereas high intakes of specific fatty acids (e.g., linoieic acid) increased risk. The cohort size and 13-year follow-up provided >90 percent power to detect a trend across quintiles of dietary intake. In 1998, among approximately 2,400 prevalent cases with diet data, study investigators addressed a secondary aim: to determine the relation of dietary factors to COPD severity during 1998-2000. COPD severity was assessed by self-report of current medications, recent symptoms, activity limitations, and health care utilization (e.g., emergency room or urgent office visits for COPD exacerbations). The rising prevalence of COPD, particularly among women, along with its high societal cost, makes COPD prevention an important public health goal.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-07; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Camargo — Brigham and Women's Hospital

REFERENCES:
- [Background] Barr RG, Somers SC, Speizer FE, Camargo CA Jr; National Asthma Education and Prevention Program (NAEPP). Patient factors and medication guideline adherence among older women with asthma. Arch Intern Med. 2002 Aug 12-26;162(15):1761-8. doi: 10.1001/archinte.162.15.1761. PMID 12153380
- [Background] Kim S, Camargo CA Jr. Sex-race differences in the relationship between obesity and asthma: the behavioral risk factor surveillance system, 2000. Ann Epidemiol. 2003 Nov;13(10):666-73. doi: 10.1016/s1047-2797(03)00054-1. PMID 14599730
- [Background] Rana JS, Mittleman MA, Sheikh J, Hu FB, Manson JE, Colditz GA, Speizer FE, Barr RG, Camargo CA Jr. Chronic obstructive pulmonary disease, asthma, and risk of type 2 diabetes in women. Diabetes Care. 2004 Oct;27(10):2478-84. doi: 10.2337/diacare.27.10.2478. PMID 15451919
- [Background] Barr RG, Wentowski CC, Grodstein F, Somers SC, Stampfer MJ, Schwartz J, Speizer FE, Camargo CA Jr. Prospective study of postmenopausal hormone use and newly diagnosed asthma and chronic obstructive pulmonary disease. Arch Intern Med. 2004 Feb 23;164(4):379-86. doi: 10.1001/archinte.164.4.379. PMID 14980988
- [Background] Griswold SK, Nordstrom CR, Clark S, Gaeta TJ, Price ML, Camargo CA Jr. Asthma exacerbations in North American adults: who are the "frequent fliers" in the emergency department? Chest. 2005 May;127(5):1579-86. doi: 10.1378/chest.127.5.1579. PMID 15888831